CLINICAL TRIAL: NCT06979830
Title: The Effects of Yoga Exercises on Body Composition, Respiratory Parameters and Functional Levels in Overweight and Obese Women: A Randomized Controlled Trial
Brief Title: The Effects of Yoga Exercises in Overweight and Obese Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, MİNE PEKESEN KURTÇA, Associate Professor, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OMU2025/87
Record Dates: First submitted 2025-04-11; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Overweight and Obese Women
Keywords: overweight; obesity; yoga; body composition; pulmonary functions; depression; anxiety
MeSH Terms: conditions — Overweight; Obesity; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- yoga exercise group (Experimental): The program will run for twelve weeks, with three sessions per week, each lasting sixty minutes, under the guidance of Physiotherapist Tuğçe BAĞCI.
  Interventions: Behavioral: yoga exercises
- control group (No Intervention): Participants in this group will not receive any exercise intervention. They will be instructed not to participate in any exercise program throughout the duration of the study.

INTERVENTIONS:
Behavioral: yoga exercises — The yoga program, based on Hatha yoga content, will be conducted in groups of 10 participants, for 12 weeks, 3 days a week, at the same time each day (12:00-13:00), and will be administered by an experienced physiotherapist (Appendix 4).
  Before starting the training program, the exercise group will be given a one-week adaptation period, during which the exercises to be performed in three sessions per week will be taught.
  Participants in the exercise group who miss sessions for various reasons will be given an additional one-week period to make up for missed sessions. Participants who miss more than four sessions will be excluded from the study.
  Participants were informed in advance about any personal items they might need before each yoga session (such as towels, tissues, etc.) and were advised to bring their own. The yoga sessions were held in the sports hall of the Artvin Çoruh Dormitory, where the required equipment for yoga (e.g., mats, blocks) was provided. The yoga program was
  Arms: yoga exercise group

SUMMARY:
Obesity has been defined by the World Health Organization (WHO) as an abnormal accumulation of fat in the body that negatively affects health and has been reported to be the most significant public health problem of the 21st century. In the late 1990s, WHO described obesity as a "global epidemic." This epidemic and its associated complications cause the death of 2.8 million adults annually. Additionally, obesity imposes a significant financial burden on countries' healthcare and social security systems. Therefore, obesity stands out as an issue that requires urgent preventive measures.

Obesity is associated with various abnormalities in respiratory functions. Changes in respiratory system mechanics due to decreased lung volumes indicate a strong link between obesity and chronic respiratory diseases. Furthermore, obesity is a risk factor for conditions such as hypertension, cardiovascular diseases, and diabetes.

Yoga is known to have numerous positive effects on health and can provide significant benefits, particularly in improving respiratory functions. Yoga is also an important tool for coping with stress, which can positively influence the respiratory system. It has been reported that yoga reduces the impact of stress on respiratory rate, promoting deep breathing and relaxation.

Some studies on the effects of yoga on obesity have not reached significant conclusions. A study comparing the effects of Vinyasa and Hatha yoga on obesity management found that neither type had a significant effect on metabolism. These studies fail to fully explain the mechanism by which yoga affects obesity due to differences in yoga styles and their lack of standardization, variations in practice durations, and the differing characteristics of study populations. Furthermore, studies on obesity and yoga often have short intervention durations (an average of 8 weeks), with most involving 60-90 minute sessions conducted 1-2 times per week.

Since longer-term studies are needed to better understand the relationship between obesity and yoga, this study aims to investigate the effects of yoga exercises on body composition, respiratory parameters, functional level, sleep quality, quality of life, and emotional state in overweight and obese women.

DETAILED DESCRIPTION:
Obesity is a preventable yet significant health burden classified as a lifestyle disease. It is defined as excessive fat accumulation in the body, reaching levels that can negatively impact health. Body mass index (BMI) is used to classify overweight and obesity. The World Health Organization (WHO) defines overweight in adults as a BMI of 25 kg/m² or higher and obesity as a BMI of 30 kg/m² or higher. The prevalence of obesity is increasing worldwide, especially in developing countries. The point prevalence rate in women (15%) is higher than in men (11%). Over the past fifty years, global obesity rates have tripled. A study determined that over 1.9 billion adults aged 18 and older were overweight, with 650 million of them classified as obese.

Obesity is a known risk factor for numerous chronic diseases, including hypertension, hyperlipidemia, type 2 diabetes, coronary heart disease, stroke, cancer, depression, and knee osteoarthritis. Since a sedentary lifestyle is one of the primary causes of obesity, regular physical activity is recommended as a treatment option for non-morbid obesity. Various studies have demonstrated a strong inverse relationship between physical activity and BMI. However, it is well known that obese individuals face challenges in increasing and maintaining physical activity levels. Therefore, there is a search for pragmatic interventions that are easy to implement and promote increased physical activity for sustainable weight loss in obese individuals.

According to the 2012 report of the National Health Statistics in the United States, the prevalence of using any complementary medicine method among adults over 18 years old was 33.2%, with yoga being one of the most frequently preferred methods. Compared to other exercises, yoga offers several advantages, such as being independent of weather conditions, requiring no financial cost, and being applicable in both indoor and outdoor settings, which has contributed to its increasing popularity and widespread adoption.

Yoga, derived from the Sanskrit word meaning "union," aims to harmonize the mind, body, and spirit. Traditional yoga consists of the eight limbs defined by Patanjali: Yamas and Niyamas (moral and ethical restraints), Asanas (postures), Pranayama (breath regulation), Pratyahara (withdrawal of senses), Dharana (concentration), Dhyana (meditation), and Samadhi (self-realization). Yoga is designed to enhance both physical and mental health, thus improving overall quality of life. Numerous studies have shown that yoga reduces stress levels and enhances general well-being. In addition to its physical health benefits, yoga positively impacts psychological health. Research suggests that yoga can improve body image and quality of life.

The current U.S. National Physical Activity Guidelines categorize yoga as a light-intensity (such as Hatha yoga) or moderate-intensity (such as Vinyasa or power yoga) physical activity, depending on the style. Additionally, yoga can function as both an aerobic and strength-based exercise, depending on the style and postures practiced. The guidelines recommend 150-300 minutes of moderate-intensity yoga per week for adults. The American College of Sports Medicine classifies yoga as a neuromotor exercise, suggesting its practice at least 2-3 times per week for 20-30 minutes per session without specifying intensity levels. Yoga has several benefits, including preventing weight gain, reducing body fat mass, and increasing lean body mass.

Mooventhan and Khode conducted a study involving 40 participants in the yoga group and 39 in the control group, where 10-minute morning yoga sessions, six days a week for two weeks, significantly reduced body weight. Similarly, Kanojia et al. found a statistically significant reduction in body weight among healthy women aged 18-20 who practiced yoga for 40 minutes, six times a week, over three menstrual cycles compared to the control group.

Yoga postures can serve as a moderate-intensity exercise for individuals with limited aerobic capacity or restricted exercise ability. While enhancing physical strength, flexibility, and endurance, yoga also improves sleep patterns. Research suggests that yoga practices can have beneficial effects on sleep disorders. Yoga promotes relaxation and reduces stress and anxiety, thereby improving sleep quality. Several scientific studies have demonstrated that yoga techniques such as Pranayama and meditation help enhance sleep quality and alleviate insomnia.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years
* Body Mass Index (BMI) ≥ 25
* Waist circumference > 88 cm
* Waist-to-hip ratio > 0.8
* Being literate, willing to participate, and signing the informed consent form
* No mental disorders
* No orthopedic or neurological conditions affecting balance
* No history of surgical operations in the last 6 months

Exclusion Criteria:

* Pregnant and breastfeeding mothers
* Participants following any diet program for obesity
* Individuals with syndromic or endocrine-related obesity
* Participants who regularly exercise
* Individuals using psychiatric medication
* Participants with a medical history that would prevent them from practicing yoga
* Participants with cardiovascular diseases that prevent exercise
* Participants with a yoga history within the last 6 months
* Individuals with any complications of obesity requiring medication, such as Type 2 diabetes or Stage 2 hypertension
* Experiencing pain over 7 on the Visual Analog Scale (VAS)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — WOMEN
Enrollment: 50 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Forced Vital Capacity (FVC) | From enrollment to the end of treatment at twelve weeks
  Spirometry is a fundamental test for assessing lung function and is essential for the evaluation and monitoring of respiratory diseases. Spirometry is a physiological test that measures the maximum effort a person can exhale and the maximum volume of air they can exhale. For the evaluation of lung function, a Care Fusion brand spirometry device will be used. Before the test, the patient's gender, age, height, and weight will be recorded in the device. The patient will be seated in a position that facilitates the required maneuvers, and nasal breathing will be prevented by placing a nose clip. After three test measurements with 95% consistency, the best value obtained will be used.
Assessment of Dynamic Balance and Functional Level (Timed Up and Go Test) | From enrollment to the end of treatment at twelve weeks"
  The test, originally called the "Timed Up & Go Test," is frequently used to measure the functional status of the lower extremities. This test also assesses individuals' ability to maintain balance during transfers and walking. In this test, individuals are asked to sit on a standard fourtyfive cm high chair with their feet flat on the ground, then stand up, walk as quickly but safely as possible for three meters, turn around at the marked point three meters away, walk back toward the chair, and sit down again. The time taken between starting and finishing the test is recorded in seconds using a stopwatch. Individuals are asked to repeat the test three times, and the average of the three trials is used for analysis.
Body Mass Index | From enrollment to the end of treatment at twelve weeks
  Weight (kg): The Tanita BIA scale device will measure the individual's body weight in kilograms. This measurement is essential for calculating other body composition parameters and assessing overall health. Height (cm): A stadiometer with an accuracy of ±0.5 cm will be used to measure the individual's height in centimeters. Accurate height measurement is fundamental for calculating body mass index (BMI) and assessing growth patterns.After completing the measurements, the dietitian will calculate the BMI by dividing weight in kilograms by the square of height in meters. BMI is a widely used indicator to assess whether an individual has a healthy body weight for a given height.
Waist Circumference | From enrollment to the end of treatment at twelve weeks
  Waist circumference will be measured at the midpoint between the lower margin of the last palpable rib and the top of the iliac crest, using a non-stretch tape measure. The individual will stand with feet close together, arms at the sides, and body weight evenly distributed. The measurement will be taken at the end of a normal expiration, ensuring the tape is horizontal and snug but not compressing the skin.
Hip Circumference | From enrollment to the end of treatment at twelve weeks
  Hip circumference will be measured around the widest portion of the buttocks, with the tape parallel to the floor. The individual will stand with feet close together, arms at the sides, and body weight evenly distributed. The measurement will be taken to the nearest 0.1 cm, ensuring the tape is snug but not compressing the skin.
Forced Expiratory Volume at One Second (FEV1) | From enrollment to the end of treatment at twelve weeks
  Spirometry is a fundamental test for assessing lung function and is essential for the evaluation and monitoring of respiratory diseases. Spirometry is a physiological test that measures the maximum effort a person can exhale and the maximum volume of air they can exhale. For the evaluation of lung function, a Care Fusion brand spirometry device will be used. Before the test, the patient's gender, age, height, and weight will be recorded in the device. The patient will be seated in a position that facilitates the required maneuvers, and nasal breathing will be prevented by placing a nose clip. After three test measurements with 95% consistency, the best value obtained will be used.
Peak Expiratory Flow (PEF) | From enrollment to the end of treatment at twelve weeks
  Spirometry is a fundamental test for assessing lung function and is essential for the evaluation and monitoring of respiratory diseases. Spirometry is a physiological test that measures the maximum effort a person can exhale and the maximum volume of air they can exhale. For the evaluation of lung function, a Care Fusion brand spirometry device will be used. Before the test, the patient's gender, age, height, and weight will be recorded in the device. The patient will be seated in a position that facilitates the required maneuvers, and nasal breathing will be prevented by placing a nose clip. After three test measurements with 95% consistency, the best value obtained will be used.
Maximum Mid-expiratory Flow 25-75% (MMEF25-75) | From enrollment to the end of treatment at twelve weeks
  Spirometry is a fundamental test for assessing lung function and is essential for the evaluation and monitoring of respiratory diseases. Spirometry is a physiological test that measures the maximum effort a person can exhale and the maximum volume of air they can exhale. For the evaluation of lung function, a Care Fusion brand spirometry device will be used. Before the test, the patient's gender, age, height, and weight will be recorded in the device. The patient will be seated in a position that facilitates the required maneuvers, and nasal breathing will be prevented by placing a nose clip. After three test measurements with 95% consistency, the best value obtained will be used.
FEV1/FVC | From enrollment to the end of treatment at twelve weeks
  Spirometry is a fundamental test for assessing lung function and is essential for the evaluation and monitoring of respiratory diseases. Spirometry is a physiological test that measures the maximum effort a person can exhale and the maximum volume of air they can exhale. For the evaluation of lung function, a Care Fusion brand spirometry device will be used. Before the test, the patient's gender, age, height, and weight will be recorded in the device. The patient will be seated in a position that facilitates the required maneuvers, and nasal breathing will be prevented by placing a nose clip. After three test measurements with 95% consistency, the best value obtained will be used.
Weight (kg) | From enrollment to the end of treatment at twelve weeks
  Weight analysis will be conducted under the supervision of a dietitian using the Tanita bioelectrical impedance analysis (BIA) scale device to measure.
Fat Percentage (%) | From enrollment to the end of treatment at twelve weeks
  Fat Percentage (%) analysis will be conducted under the supervision of a dietitian using the Tanita bioelectrical impedance analysis (BIA) scale device to measure.
Height (cm) | From enrollment to the end of treatment at twelve weeks
  For height measurement (cm), a stadiometer (±0.5 cm) will be used.
Fat Mass (kg) | From enrollment to the end of treatment at twelve weeks
  Fat Mass (kg) analysis will be conducted under the supervision of a dietitian using the Tanita bioelectrical impedance analysis (BIA) scale device to measure.
Muscle Mass (kg) | From enrollment to the end of treatment at twelve weeks
  Muscle Mass (kg) analysis will be conducted under the supervision of a dietitian using the Tanita bioelectrical impedance analysis (BIA) scale device to measure.
Muscle Percentage (%) | From enrollment to the end of treatment at twelve weeks
  Muscle percentage (%) analysis will be conducted under the supervision of a dietitian using the Tanita bioelectrical impedance analysis (BIA) scale device to measure.

SECONDARY OUTCOMES:
Assessment of Quality of Life (Short Form-36) | From enrollment to the end of treatment at twelve weeks"
  In general terms, quality of life is defined as an individual's perception of their situation in life, in the context of their cultural values, expectations, and desires. The Short Form-36 is a generic, broad-scale measurement tool within quality of life scales. It was developed and made available by the RAND Corporation. The reliability and validity of the Turkish version were assessed by Koçyiğit and colleagues. The survey is divided into eight subcategories: social functioning, physical functioning, emotional functioning, physical role limitations, general health status, mental health status, pain, and vitality (energy), and consists of thirty-six questions. Scoring is done on a scale from zero to one hundred, where zero indicates very poor health status and one hundred indicates no health problems.
Assessment of Sleep Quality (Pittsburgh Sleep Quality Index - PSQI) | From enrollment to the end of treatment at twelve weeks"
  The Pittsburgh Sleep Quality Index (PSQI) was developed by Buysse et al. and adapted into Turkish by Ağargün et al. The PSQI is a nineteen-item self-report scale that evaluates sleep quality and disturbances over the past month. It consists of twenty-four questions, nineteen of which are self-report items, while five questions are answered by a bed partner or roommate. The eighteen scored questions of the scale are divided into seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, sleep medication use, and daytime dysfunction. Each component is scored on a zero to three scale. The total score of the scale is derived from the sum of the seven components. The total score ranges from zero to twenty-one. A total score greater than five indicates poor sleep quality.
Assessment of Emotional Status (Beck Depression Inventory (BDI)) | From enrollment to the end of treatment at twelve weeks"
  The BAI was developed by Aaron Beck. It consists of twenty-one questions related to common anxiety symptoms such as sweating, trembling, fear, and distress, and asks how the individual has felt during the past week, including the current day. The aim is to measure the anxiety levels present in individuals. In this scale, each item has four options, and the scoring ranges from zero to three (zero points for "Not at all"; one point for "Mild level (didn't affect me)"; two points for "Moderate level (it was unpleasant but bearable)"; three points for "Severe level (I had difficulty bearing it)"). The total score obtained from the answers ranges from zero to sixty-three. At the end of the test, the scores are totaled. The categorization is as follows: eight to fifteen points: mild anxiety symptoms; sixteen to twenty-five points: moderate anxiety symptoms; twenty-six to sixty-three points: severe anxiety symptoms. The internal consistency reliability was found to be eighty-six.
Assessment of Emotional Status (Beck Anxiety Inventory (BAI)) | From enrollment to the end of treatment at twelve weeks"
  The BAI, developed by Aaron Beck, consists of twenty-one questions assessing common anxiety symptoms such as sweating, trembling, fear, and distress. It evaluates how individuals have felt over the past week, including the current day. Each item has four response options, scored from zero to three. The total score ranges from zero to sixty-three. Anxiety levels are categorized as mild (eight to fifteen), moderate (sixteen to twenty-five), and severe (twenty-six to sixty-three). The reliability coefficient of the scale in Turkey was reported as Cronbach's alpha = 0.92.

REFERENCES:
- [Background] Ulusoy, M., Sahin, N. H., & Erkmen, H. (1998). Turkish version of the Beck Anxiety Inventory: psychometric properties. Journal of cognitive psychotherapy, 12(2), 163.
- [Background] Telles S, Sharma SK, Singh A, Kala N, Upadhyay V, Arya J, Balkrishna A. Quality of Life in Yoga Experienced and Yoga Naive Asian Indian Adults with Obesity. J Obes. 2019 Apr 30;2019:9895074. doi: 10.1155/2019/9895074. eCollection 2019. PMID 31183215
- [Background] Shohani M, Badfar G, Nasirkandy MP, Kaikhavani S, Rahmati S, Modmeli Y, Soleymani A, Azami M. The Effect of Yoga on Stress, Anxiety, and Depression in Women. Int J Prev Med. 2018 Feb 21;9:21. doi: 10.4103/ijpvm.IJPVM_242_16. eCollection 2018. PMID 29541436
- [Background] Panwar, S. H. E. E. T. A. L., Chourishi, A. S. H. U. T. O. S. H., & Makwana, J. A. Y. A. N. T. (2012). Effect of pranayama (yoga) on pulmonary function test of young healthy students. Int J Pharma Bio Sci, 3(4), 12-6.
- [Background] Kargün, M., Togo, O. T., Biner, M., & Pala, A. (2016). Üniversite öğrencilerinin fiziksel aktivite düzeylerinin incelenmesi. Marmara Üniversitesi Spor Bilimleri Dergisi, 1(1), 61-72.
- [Background] Hisli, N. (1989). Beck depresyon envanterinin universite ogrencileri icin gecerliligi, guvenilirligi.(A reliability and validity study of Beck Depression Inventory in a university student sample). J. Psychol., 7, 3-13.
- [Background] Gündede, E. (2018). Serebral palsili çocukların fonksiyonelliği ile ebeveynlerinin bakım yükü, aktivite düzeyi, yaşam kalitesi ve psikolojik durumu arasındaki ilişki. Okan Üniversitesi, İstanbul.
- [Background] Cramer H, Thoms MS, Anheyer D, Lauche R, Dobos G. Yoga in Women With Abdominal Obesityߞa Randomized Controlled Trial. Dtsch Arztebl Int. 2016 Sep 30;113(39):645-652. doi: 10.3238/arztebl.2016.0645. PMID 27776622
- [Background] Asiah ASS, Norhayati MN, Muhammad J, Muhamad R. Effect of yoga on anthropometry, quality of life, and lipid profile in patients with obesity and central obesity: A systematic review and meta-analysis. Complement Ther Med. 2023 Sep;76:102959. doi: 10.1016/j.ctim.2023.102959. Epub 2023 Jun 24. PMID 37356673